CLINICAL TRIAL: NCT03787329
Title: The Effect of Autologous Bone Marrow Concentration Combined With Core Decompression for Avascular Necrosis of Femoral Head
Brief Title: Autologous Bone Marrow Concentration for Avascular Necrosis of Femoral Head
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Superintendent, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Other Study IDs: RD-106057
Record Dates: First submitted 2018-12-22; First posted 2018-12-26 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Avascular Necrosis of Femur; Bone Marrow
Keywords: Femur Head Necrosis; Mesenchymal Stromal Cells; Bone Marrow
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone marrow concentration group: The patients receive core decompression surgery with bone marrow concentration.
  Interventions: Other: Core decompression surgery with bone marrow concentration
- Historical control group: The previous age-, gender-, and stage-matched patients who received core decompression surgery only.
  Interventions: Other: Core decompression surgery

INTERVENTIONS:
Other: Core decompression surgery with bone marrow concentration — Core decompression surgery with bone marrow concentration
  Groups: Bone marrow concentration group
Other: Core decompression surgery — Core decompression surgery only
  Groups: Historical control group

SUMMARY:
This study aims to evaluate the effect of bone marrow concentration on avascular necrosis of femur head by comparing clinical and imaging outcomes between patients receiving core decompression surgery with intraoperative bone marrow concentration and those receiving core decompression surgery only.

DETAILED DESCRIPTION:
Avascular necrosis (AVN) of femoral head is a progressive disease that predominantly affects younger patients. Although the exact pathophysiology of AVN has not yet to be elucidated, the disease is characterized by a vascular insult to the blood supply of the femoral head, which can lead to collapse of the femoral head and subsequent degenerative changes. Mesenchymal stem cells (MSCs) are pluripotent cells that can differentiate into multiple mesenchymal tissues, including tenocytes, chondrocytes and osteoblasts, as well as being a source of multiple growth factors to establish an environment conducive to soft and hard tissue regeneration. As bone marrow concentration has high concentration of mesenchymal stem cells, several studies have applied the autologous bone marrow concentration in halting the progression of AVN of femoral head. However, a higher level of evidence for its use on patients suffering from femoral head avascular necrosis has not been reported. This clinical trial will evaluate and compare the eligible patients who undertake core decompression surgery plus intraoperative bone marrow concentration with those who received core decompression surgery only. All patients will be followed for one year and clinical and imaging outcomes will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 60 years
* With diagnosis of avascular necrosis of femoral head, Stage I - Stage III

Exclusion Criteria:

* With diagnosis of avascular necrosis of femoral head, Stage VI - Stage VI
* With prior history of hip surgery
* With current or prior history of trauma or infection at hip
* Platelet count < 50,000/µL
* With current diagnosis of coagulopathy
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: consecutive eligible patients who underwent core decompression combined with autologous bone marrow stem cells treatment for avascular necrosis of the femoral head
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
3-month postoperative hip function evaluated by Harris Hip Score | 3-month postoperative
  Hip function is evaluated using Harris Hip score. The survey has 10 question items and scores range from 0-100 with higher scores representing less dysfunction and better outcomes.

SECONDARY OUTCOMES:
6-month postoperative hip function evaluated by Harris Hip Score | 6-month postoperative
  Hip function is evaluated using Harris Hip Score. The survey has 10 question items and scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
12-month postoperative hip function evaluated by Harris Hip Score | 12-month postoperative
  Hip function is evaluated using Harris Hip Score. The survey has 10 question items and scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
3-month postoperative degree of collapse evaluated by plain radiograph | 3-month postoperative
  Degree of collapse is evaluated by plain radiograph
6-month postoperative degree of collapse evaluated by plain radiograph | 6-month postoperative
  Degree of collapse is evaluated by plain radiograph
12-month postoperative degree of collapse evaluated by plain radiograph | 12-month postoperative
  Degree of collapse is evaluated by plain radiograph
6-month postoperative degree of collapse evaluated by MRI | 6-month postoperative
  Degree of collapse is evaluated by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No